CLINICAL TRIAL: NCT04610021
Title: Prospective Analysis of the i-FactorTM Bone Graft on the Fusion Rate and Quality of Life of Patients With Adult Spine Deformity
Brief Title: Prospective i-FactorTM Analysis Fusion Rate and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Asistencial Universitario de León Urgencias (Other)
Responsible Party: Principal Investigator, Manuel Fernández González, Jefe de Servicio, Complejo Asistencial Universitario de León Urgencias
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: CAULE-IFACTOR
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Spinal Deformity; Bone Graft; Fusion Rate; Quality of Life
Keywords: Adult Spinal deformity; Bone graft; Fusion rate; Quality of life; Spinal Surgery; Functional limitations

STUDY DESIGN:
Intervention Model Description: prospective randomized with intervention study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): Control group: autologous bone + bench bone
- i-Factor (Experimental): I-Factor group: autologous bone + bench bone + i-Factor™ bone graft
  Interventions: Biological: i-FactorTM Bone graft

INTERVENTIONS:
Biological: i-FactorTM Bone graft — In the i-Factor ™ group it will be placed longitudinally in the intertransverse area. Likewise, in both groups, only autologous and bench bone will be placed in the intersomatic cages. The vertebrae where the i-Factor ™ is placed will be noted on the data collection sheet.
  Arms: i-Factor

SUMMARY:
Adult spinal deformity surgery is a complex procedure that involves many risks and complications. Bone grafts and bone substitutes are essential to achieve fusion and manage stability in spinal surgery.

Autologous bone has been considered the "gold-standard" for obtaining a spinal fusion. However, the source from which to obtain it is limited. Furthermore, the problems of bone quality in patients with osteoporosis and the morbidity have forced the orthopedic community to seek other options.

I-Factor ™ Bone Graft (Cerapedics, Inc., Westminster, CO) is a compound formed by peptide P-15 bound to an anorganic bone mineral of bovine origin that is composed of porous and smooth hydroxyapatite (ABM) particles.

In the literature there are no articles which identify bone formation with the i-Factor ™ graft in more than 4 instrumented levels, therefore the development of this study will allow assessing the fusion rate and quality of life of patients, which could lead to an improvement in the management and decision-making of surgical procedures, as well as better control of healthcare spending

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age.
* Patients diagnosed with adult deformity, whether due to scoliosis, imbalance, thoracolumbar curves, etc. In which the minimum number of levels to be instrumented is 5, that is, 4 intervertebral discs.
* Patients who provide their informed consent in writing. (In the event that the patient's circumstances do not allow him to grant consent, this may be provided by the legal representative).
* Present radiological tests, computed tomography and / or magnetic resonance imaging prior to surgery.
* The implants used in the surgery are Cobalt Chrome bars and Titanium screws and interbody cages.

Exclusion Criteria:

* Patients who are expected to be unavailable for follow-up.
* Patients with mental disabilities that make it difficult for them to fill in the questionnaires.
* Patients who have had other types of implants placed, other than Cobalt Chrome bars and Titanium screws and interbody cages.
* Patients who are going to have cemented and / or expansive screws, Peek boxes or another type of material other than Titanium.
* Underlying neurological or neuromuscular disease.
* Underlying inflammatory or tumor disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Fusion rate | 2 years
  The success of the fusion at 12 and 24 months will be determined by a specialized radiologist by the evidence in the CT scan of trabecular bone bridges between the inter-transverse areas of the vertebral bodies and the absence of radiolucency adjacent to the implants.
Minimal Clinically Important Difference (MCID) | 2 years
  Minimal clinically important difference is defined a smallest clinical change that is important to the patient.
Short Form Health Survey-12 General Quality of life questionnaire | 2 years
  The questions that follow ask what you think about your health. Your answers will allow you to know how you are and to what extent you are able to do your usual activities.
  Patients improve when the puntuation is more than 50.
Owestry disability index | 2 years
  Disability index questionnaire
  Maximun value=100 Minimun value=0
  Patients improve when this index is arround 0
VISUAL ANALOGUE SCALE | 2 years
  Is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  Maximun value=10 Minimun value=0
  Patients improve when this index is arround 0
Scoliosis Research Society (SRS-22) | 2 years
  Scoliosis reseach society questionnaire
  22 questions 5 options Dimensions Pain Function Selfimage Mental Health Satrisfaction
  Puntuation for item and test: 1(worse) - 5(better)

CONTACTS AND LOCATIONS:
Locations (1):
- CAULE, León, Spain